CLINICAL TRIAL: NCT03563690
Title: Different Kinds of Acupuncture Treatment for Knee Osteoarthritis：a Multicentre Randomised Controlled Trial
Brief Title: Different Kinds of Acupuncture Treatment for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); Jiaxing TCM Hospital (Unknown); Zhejiang Provincial Hospital of TCM (Other); Zhejiang Hospital (Other); Red Cross Hospital, Hangzhou, China (Other); Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018ZY008-KOA
Record Dates: First submitted 2018-05-17; First posted 2018-06-20 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
Keywords: KOA; Acupuncture treatment; Multi-center RCT
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Acupuncture group (Experimental): When recruited from six centers,the participant will be randomized to six groups .In acupuncture group participant will receive four-week acupuncture treatment(three times a week )continuously for 4 weeks,12 treatments in total. The follow-up period is six months.
  Interventions: Other: treatment1
- Electro-acupuncture group (Experimental): When recruited from six centers,the participant will be randomized to six groups. In this group participant receive four-week electro-acupuncture treatment(three times a week )continuously for 4 weeks,12 treatments in total. The follow-up period is six months.
  Interventions: Other: treatment2
- Moxibustion group (Experimental): When recruited from six centers,the participant will be randomized to six groups. In this group participant receive four-week moxibustion treatment (three times a week )continuously for 4 weeks,12 treatments in total. The follow-up period is six months.
  Interventions: Other: treatment3
- Warm-needling group (Experimental): When recruited from six centers,the participant will be randomized to six groups. In this group participant receive four-week warm-needling treatment (three times a week )continuously for 4 weeks,12 treatments in total. The follow-up period is six months.
  Interventions: Other: treatment4
- Sham-needle group (Sham Comparator): When recruited from six centers,the participant will be randomized to six groups.In this group participant receive four-week sham acupuncture treatment (three times a week )continuously for 4 weeks,12 treatments in total. The follow-up period is six months.
  Interventions: Other: treatment5
- Celebrex group (Active Comparator): When recruited from six centers,the participant will be randomized to six groups . In this group participant will receive Celebrex (Celebrex, Capsules, Pfizer Pharmaceuticals Ltd)treatment, which will be applied 1 time daily(one time oral 0.2g) for 4 weeks. The follow-up period is six months.
  Interventions: Drug: Celebrex

INTERVENTIONS:
Other: treatment1 — 1. Acupoints：Liangqiu（ST34）,Xuehai（SP10）,Neixiyan（EX-LE4）,Dubi(ST35),Yanglingquan (GB34)and Yinlingquan (SP9)
  2. operation: the needles will be manipulated using techniques including lifting, thrusting, twisting, and rotating, until De Qi is achieved for 30 minutes.
  Arms: Acupuncture group
Other: treatment2 — 1. Acupoints：Needling points are the same to the above group
  2. operation: The electrode will be connected Neixiyan (EX-LE4) and Dubi (ST35) and electrode wire will be connected to the electro-acupuncture apparatus using dilatational wave with a frequency of 2/100 Hz, the current intensity is within participants'tolerance, for 30 minutes.
  Arms: Electro-acupuncture group
Other: treatment3 — 1. Acupoints：treating points are the same to the above group
  2. Operation: During treatment, participants will choose to sit with knee buckling natural 90 degrees ,with the affected knee(s) exposed. Mild moxibustion are applied at the distance of 2-3 cm away from the skin of both the Neixiyan (EX-LE4) and Dubi (ST35) for 30 minutes.
  Arms: Moxibustion group
Other: treatment4 — 1. Acupoints：Needling points are the same to the above group
  2. Operation: Warm-needling acupuncture are applied at both Neixiyan (EX-LE4) and Dubi (ST35). That is to insert one zhuang(about 2cm)of Huai Qing Ai on the top of the needle, and burn the moxa at the lower end ,each acupoint applied 2 Zhuang for 30 minutes.
  Arms: Warm-needling group
Other: treatment5 — 1. points：Sham Liangqiu（ST34）,Sham Xuehai(SP10), Sham Neixiyan(EX-LE4), Sham Yanglingquan(GB34),Sham Yinlingquan (SP9)
  2. Operation: Sham acupuncture with non-meridian and non-acupoint needling method, respectively acupuncture 1cm away lateral to the above sham acupoints with a 0.18 * 25mm single-use needle with the depth of 1-2mm.
  Arms: Sham-needle group
Drug: Celebrex — Drug: Celebrex (Celebrex, Capsules, Pfizer Pharmaceuticals Ltd), which will be applied 1 time daily( taken 0.2g one time orally ) Time of treatment :4 weeks Other Name: celecoxib
  Arms: Celebrex group

SUMMARY:
Knee osteoarthritis (KOA) a chronic disease with symptoms of persistent pain or rest pain , joint stiffness, numbness, limitation of activity and even disability, with significant associated costs and effects on individuals' life quality. Acupuncture as an approach for the management of chronic pain, is receiving increasing recognition from both the public and professionals. The aim of this study is to indicate the effects of three commonly used acupuncture treatments for KOA.

DETAILED DESCRIPTION:
360 subjects with KOA recruited from six centers will be randomized to six groups ,and receive four-week acupuncture, Electro-acupuncture, Moxibustion ,Warm-needling ,sham-needle, celebrex treatment. The primary outcomes are Visual Analogue Scale (VAS) and WOMAC function score.The Secondary outcomes are WOMAC pain score, WOMAC stiffness score,the Physical Activity Scale of the Elderly (PASE),knee joint swelling measurement and WHO-BREF life quality scale.The follow-up period is six months. This study will be a rigorous,randomized, sham and drug controlled trial focusing on using different kinds of acupuncture treatment for treating KOA.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Clinical Classification Criteria for Osteoarthritis of the Knee, diagnosed by specialist.
2. Aged 40-75 years old;
3. History of chronic knee pain for more than 3 months, and complain of knee pain on most days of the past month;
4. Kellgren and Lawrence Grades 1-3;
5. With related knee pain in one or both knees rated > 4 cm on a 10 cm Visual Analog Scale(VAS) (VAS:0 to 10)
6. Who volunteer to participate and sign the consent form .

Exclusion Criteria:

1. Knee osteoarthritis patients with gout, infection, tumor, autoimmune diseases, trauma or other causes of knee pain or knee deformities;
2. Patients who have local skin damage, poor skin conditions or coagulant dysfunction and patients who are not suitable for acupuncture;
3. Patients who are accompanied with serious medical problems or mental disorders, cognitive dysfunction，disorders of shallow sensation or who cannot cooperate with the treatment;
4. Patients who have received acupuncture or needle knife in the past month;
5. Other patients who are not suitable for acupuncture treatment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score change | baseline,2 weeks, 4 weeks ,3 months,6months
  Intensity of pain range (lately 3 days' average): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain.
WOMAC function change | baseline,2 weeks,4 weeks ,3 months,6months
  The WOMAC function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.

SECONDARY OUTCOMES:
WOMAC pain change | baseline,2 weeks,4weeks ,3 months,6months
  The WOMAC pain subscale referred to the patient's pain. It was comprised of 5 items, with each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst pain condition. An overall score range of 0 (minimum) to 20 (maximum), with higher scores indicating worse physical function.
WOMAC stiffness change | baseline,2 weeks,4 weeks ,3 months,6months
  The WOMAC stiffness subscale was comprised of 2 questions regarding the degree of stiffness experienced in the study knee. The WOMAC stiffness subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse stiffness. An overall score range of 0 (minimum) to 8 (maximum), with higher scores indicating more stiffness.
PASE change | baseline,2 weeks,4 weeks ,3 months,6months
  Physical Activity Scale for the Elderly was comprised of 36 questions regarding physical activity of elderly's house hold,leisure,work performance with different score weight.The higher scores indicating better physical activity.
Quality of life change | baseline,2 weeks,4 weeks ,3 months,6months
  WHO-BREF 36-Item Form assessing quality of life was comprised of 26 items which measured the following broad domains: physical health, psychological health, social relationships, and environment.With higher scores indicating better quality of life.
Knee swelling measurement change | baseline,2 weeks, 4 weeks ,3 months,6months
  0-3 score indicating swelling and average Knee circumference of three times.
Expectancy questionnaires | baseline
  Expectancy questionnaires were comprised of two brief items assessing the expectancy of the patients about acupuncture(or/and)moxibustion.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D,M.D, Principal Investigator — Zhejiang CMU
Locations (1):
- The third affiliated hospital of Zhejiang CMU, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Gelber AC. Conventional medical therapy for osteoarthritis: current state of the evidence. Curr Opin Rheumatol. 2015 May;27(3):312-7. doi: 10.1097/BOR.0000000000000164. PMID 25784383
- [Result] Holla JF, van der Leeden M, Knol DL, Roorda LD, Hilberdink WK, Lems WF, Steultjens MP, Dekker J. Predictors and outcome of pain-related avoidance of activities in persons with early symptomatic knee osteoarthritis: a five-year followup study. Arthritis Care Res (Hoboken). 2015 Jan;67(1):48-57. doi: 10.1002/acr.22381. PMID 24905958
- [Result] WHO Scientific Group on the Burden of Musculoskeletal Conditions at the Start of the New Millennium. The burden of musculoskeletal conditions at the start of the new millennium. World Health Organ Tech Rep Ser. 2003;919:i-x, 1-218, back cover. PMID 14679827
- [Result] Xiang YJ, Dai SM. Prevalence of rheumatic diseases and disability in China. Rheumatol Int. 2009 Mar;29(5):481-90. doi: 10.1007/s00296-008-0809-z. Epub 2008 Dec 6. PMID 19066899
- [Result] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Derived] Sun J, Liang Y, Luo KT, Shao XM, Tu MQ, Wu XT, Liu F, Li XW, Chen YD, Zhang QF, Ji CH, Li RR, Li XY, Xu F, Fang JQ. Efficacy of Different Acupuncture Techniques for Pain and Dysfunction in Patients with Knee Osteoarthritis: A Randomized Controlled Trial. Pain Ther. 2025 Apr;14(2):737-751. doi: 10.1007/s40122-025-00713-x. Epub 2025 Feb 17. PMID 39961986
- [Derived] Zhang Q, Fang J, Chen L, Wu J, Ni J, Liu F, Sun J. Different kinds of acupuncture treatments for knee osteoarthritis: a multicentre, randomized controlled trial. Trials. 2020 Mar 14;21(1):264. doi: 10.1186/s13063-019-4034-8. PMID 32171318
- See also: Related Info — http://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=1&SID=7DIY5PMzIE2Bx3pNLBh&page=1&doc=1
- See also: Related Info — http://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=5&SID=7DIY5PMzIE2Bx3pNLBh&page=1&doc=1
- See also: Related Info — http://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=6&SID=7DIY5PMzIE2Bx3pNLBh&page=1&doc=9
- See also: Related Info — http://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=8&SID=7DIY5PMzIE2Bx3pNLBh&page=2&doc=85
- See also: Related Info — http://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=11&SID=7DIY5PMzIE2Bx3pNLBh&page=1&doc=2
- See also: Related Info — http://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=14&SID=7DIY5PMzIE2Bx3pNLBh&page=2&doc=69

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03563690/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03563690/ICF_001.pdf